CLINICAL TRIAL: NCT04983654
Title: Functional and Mechanistic Characterization of Limb Ulcers in Patients With Sickle Cell Disease
Acronym: DrepanO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_0305; 2021-A01605-36 (Other: ID-RCB)
Record Dates: First submitted 2021-07-13; First posted 2021-07-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ulcer; Anemia; Sickle Cell Disease
Keywords: limb ulcers; sickle cell disease; microcirculation; cytokine; wound fluid
MeSH Terms: conditions — Ulcer; Anemia; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with limb ulcer (Experimental): Patients with sickle cell disease and suffering from limb ulcer
  Interventions: Diagnostic Test: patients with limb ulcers
- Patients without limb ulcer (Experimental): Patients with sickle cell disease without any limb ulcer
  Interventions: Diagnostic Test: For patients without limb ulcers

INTERVENTIONS:
Diagnostic Test: patients with limb ulcers — For patients with limb ulcers : at inclusion visit and after healing or at 6 months if ulcer does not heal:
  * Microvascular analysis (laser doppler, TcPO2),
  * Neurological analysis ( sensitivity testing with thermal and mechanical test),
  * Analysis of physical characteristics of red blood cells and inflammatory marks,
  * Analysis of cytokine and metalloproteases in the wound fluid,
  * Assessment of healing according usual treatment
  Arms: Patients with limb ulcer
Diagnostic Test: For patients without limb ulcers — For patients without limb ulcers : at inclusion visit only
  * Microvascular analysis (laser doppler, TcPO2),
  * Neurological analysis (sensitivity testing with thermal and mechanical test),
  * Analysis of physical characteristics of red blood cells and inflammatory marks
  Arms: Patients without limb ulcer

SUMMARY:
Sickle Cell Disease is the most frequent genetic disease in the world (representing one birth over 1900, in France). The polymerization of the abnormal hemoglobin (i.e., HbS) when deoxygenated is at the origin of a mechanical distortion of red blood cells (RBC) into a crescent-like shape. Sickled RBCs are very fragile and rigid, which lead patients to have severe anemia and to develop frequent and repeated painful vaso-occlusive crises. Furthermore, the repetition of sickling-unsickling cycles causes irreversible damages to the RBCs, which shorten their half-life. Accumulation of free hemoglobin and heme in the plasma is involved in blood vessels lesions in both the macro- and micro- circulation.

The resulting vascular dysfunction could explain why limb ulcers are 10 fold more frequent in patients with sickle cell disease compared to the general population and may happen at a younger age. Limb ulcers induce significant morbidity (delay of healing between 9 and 26 weeks in the french cohort), and are associated to significant pain (needing opioid pain-killer) and increase the risk of infection. Cost of care is also increased. Moreover, ulcers induce missed school and work days.

Data on cutaneous microcirculation and ulcers physiopathology in patients with sickle cell disease are scarce. We want to realise a microcirculatory and neurological functional study of patients with with and without ulcers and a characterization of biomarkers present in the blood or in the wound fluid which can participate to ulcers physiopathology.

To ensure healing, adapted therapeutics are essential. Several strategies are proposed such as: lifestyle measures (venous compression, lower limb elevation, rest), dressings, hyperbaric oxygenotherapy (also used in diabetic ulcers). The project is devoted to study the mechanisms involved in leg ulcers and the effects of therapeutical/behavioral strategies.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease (homozygous SS or Sb0)
* Age ≥ 18 years old
* Consent patients
* Social regimen

Exclusion Criteria:

* tutela or curatella
* Vaso occlusive crisis < 1 month

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Alteration of cutaneous microvascular function and peripheral sensorial neurological function in patients with limb ulcers | Day 1
  Cutaneous microvascular function is assessed with :
  * laser Doppler Including measurement of blood pressure before and after testing, heart rate before and after testing, cutaneous temperature, values of laser Doppler before and after vasodilatation with acetylcholine, deionized water, local heating (42°C)
  * TcPO2 on the first intermetatarsal space and bordering ulcer Peripheral sensorial neurological function is assessed with Von Frey monofilament, hot (50°C)/cold (4°C) test, pic-touch test and pallesthesia.

SECONDARY OUTCOMES:
Modification of hemorheological red blood cells characteristics between patients with and without ulcers | Day 1
  Analysis of hemorheological characteristics in the 2 arms after blood test with blood viscosity and RBC rheological measurements (deformability/aggregation)
Analysis of the composition of the wound fluid | Day 1
  Analysis of metalloproteases (MMP-8 and MMP-9) and inflammatory markers (TNF-alpha, Il-6, Il1-beta, VCAM 1, P-selectin) in the wound fluid
Compare pro inflammatory markers in the blood between patients with and without ulcers | At initial visit
  Analysis of inflammatory markers in the blood and comparison between the 2 arms
Assessment of healing | through study completion, an average of 6 months
  Delay of granulation tissue appearance, delay of healing according treatment used
Compare microcirculation, pro inflammatory marker in the wound fluid and in the blood and hemorheological characteristics after usual treatment to obtain healing | through study completion, an average of 6 months
  Compare results (previously described) in the group of patients with ulcers, between initial and second visit

CONTACTS AND LOCATIONS:
Overall Officials: Judith CATELLA, Dr, Principal Investigator — Service de Médecine Interne
Locations (1):
- Groupement Hospitalier Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Catella J, Turpin E, Connes P, Nader E, Carin R, Martin M, Rezigue H, Nougier C, Dargaud Y, Josset-Lamaugarny A, Dugrain J, Marano M, Leuci A, Boisson C, Renoux C, Joly P, Poutrel S, Hot A, Guillot N, Fromy B. Impaired microvascular function in patients with sickle cell anemia and leg ulcers improved with healing. Br J Haematol. 2024 Dec;205(6):2459-2469. doi: 10.1111/bjh.19785. Epub 2024 Sep 24. PMID 39318045